CLINICAL TRIAL: NCT04081545
Title: The Effect of an Opioid-free Anesthetic on Post-operative Opioid Consumption After Laparoscopic Bariatric Surgery: a Prospective, Single-blinded, Randomized Controlled Trial
Brief Title: Effect of Opioid Free Anesthetic on Post-Operative Opioid Consumption After Laparoscopic Bariatric Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Christine Oryhan (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Sponsor-Investigator, Christine Oryhan, Anesthesiologist and Pain Medicine Physician, Benaroya Research Institute
Organization: Benaroya Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CRP19060
Record Dates: First submitted 2019-08-28; First posted 2019-09-09 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use, Unspecified; Bariatric Surgery Candidate; Anesthesia
Keywords: Opioid Free Anesthesia; Bariatric Surgery; Non-Opioid Anesthesia; Ketamine; Dexmedetomidine; Lidocaine
MeSH Terms: interventions — Analgesics, Non-Narcotic

STUDY DESIGN:
Intervention Model Description: The investigators plan to enroll 196 subjects at Virginia Mason Medical Center that are undergoing laparoscopic bariatric surgery. Subjects who volunteer to be involved in the study will be randomized to either the opioid free or traditional anesthetic arm, with a computer generated arm assignment. Subjects will be blinded to the assigned arm. Group A will receive a traditional opioid restrictive general anesthetic and group B will receive an opioid-free anesthetic technique.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Goup A- Opioid-based regimen (Active Comparator): Preop - Multimodals unless contraindicated
  Induction
  * Fentanyl (50mcg IV)
  * Lidocaine 1.5mg/kg IV bolus using IBW (Ideal body weight)
  * Propofol 2-3mg/kg IV bolus
  * Neuromuscular blockade per Anesthesiology team discretion
  Maintenance
  * Sevoflurane
  * Neuromuscular blockade at discretion of anesthesiology team
  * May use fentanyl to treat SBP or HR > 20% of baseline
  Emergence
  * Neuromuscular reversal, dosed according to Virginia Mason protocol
  * May titrate fentanyl per anesthesiology team throughout the case.
  * Patient extubated and brought to PACU
  PACU opioid orders per anesthesiology team
  Post-operative Nausea/Vomiting Prophylaxis
  -4mg dexamethasone, 1mg haloperidol, scopolamine patch
  Interventions: Drug: Opioid Anesthetics
- Experimental Group B- Opioid-free regimen (Experimental): Preop - Multimodals unless contraindicated
  Induction
  * Dexmedetomidine 1mcg/kg IV bolus over 10 minutes using IBW
  * Lidocaine 1.5mg/kg IV bolus using IBW
  * Propofol 2-3mg/kg IV bolus
  * Neuromuscular blockade per Anesthesiology team discretion
  * Ketamine 0.5mg/kg IV bolus (based on IBW)
  Maintenance
  * Sevoflurane
  * Dexmedetomidine 0.4 mcg/kg/hr IV infusion using IBW (may titrate based on patient response between 0.3-0.5mcg/kg/hr)
  * Lidocaine 2mg/kg/hr IV infusion using IBW
  * May use esmolol as needed to treat SBP or HR > 20% of baseline
  * Neuromuscular blockade at the discretion of anesthesiology team
  Emergence
  * Dexmedetomidine infusion turned off during laparoscopic desufflation
  * Lidocaine infusion turned off at skin closure
  * Neuromuscular reversal, dosed according to VM protocol
  * Pt extubated and brought to PACU
  * PACU opioid orders per anesthesiology team
  Post-operative Nausea/Vomiting Prophylaxis
  -4mg dexamethasone, 1mg haloperidol, scopolamine patch
  Interventions: Drug: Non Opioid Analgesics

INTERVENTIONS:
Drug: Opioid Anesthetics — see arm/group description
  Other Names: Opioid-based regimen
  Arms: Control Goup A- Opioid-based regimen
Drug: Non Opioid Analgesics — see arm/group description
  Other Names: Opioid-free regimen
  Arms: Experimental Group B- Opioid-free regimen

SUMMARY:
A comparison of post-operative opioid use in laparoscopic bariatric surgery patients receiving opioid or opioid-free anesthesia.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-blinded, randomized controlled trial comparing the effect of an opioid-free general anesthetic versus a traditional anesthetic with a restricted quantity of opioid on postoperative opioid consumption following laparoscopic bariatric surgery. The study population will be composed of 196 subjects undergoing laparoscopic bariatric surgery at Virginia Mason Medical center randomized into two groups. The control group will receive a traditional opioid restrictive general anesthetic. The study group will receive an opioid-free anesthetic technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective laparoscopic bariatric surgery (i.e. laparoscopic roux-en-Y gastric bypass, laparoscopic sleeve gastrectomy) able to provide informed consent

Exclusion Criteria:

* Any opioid use within 4 weeks prior to surgery
* Chronic antiemetic use
* Conversion of laparoscopic to open surgery
* Patients unable to provide post-operative pain scores
* Pregnant or lactating patients
* Patients under 18 years of age
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Oryhan, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Goup A- Opioid-based Regimen: Preop - Multimodals unless contraindicated
  Induction
  * Fentanyl (50mcg IV)
  * Lidocaine 1.5mg/kg IV bolus using IBW (Ideal body weight)
  * Propofol 2-3mg/kg IV bolus
  * Neuromuscular blockade per Anesthesiology team discretion
  Maintenance
  * Sevoflurane
  * Neuromuscular blockade at discretion of anesthesiology team
  * May use fentanyl to treat SBP or HR > 20% of baseline
  Emergence
  * Neuromuscular reversal, dosed according to Virginia Mason protocol
  * May titrate fentanyl per anesthesiology team throughout the case.
  * Patient extubated and brought to PACU
  PACU opioid orders per anesthesiology team
  Post-operative Nausea/Vomiting Prophylaxis
  -4mg dexamethasone, 1mg haloperidol, scopolamine patch
  Opioid Anesthetics: see arm/group description
- Experimental Group B- Opioid-free Regimen: Preop - Multimodals unless contraindicated
  Induction
  * Dexmedetomidine 1mcg/kg IV bolus over 10 minutes using IBW
  * Lidocaine 1.5mg/kg IV bolus using IBW
  * Propofol 2-3mg/kg IV bolus
  * Neuromuscular blockade per Anesthesiology team discretion
  * Ketamine 0.5mg/kg IV bolus (based on IBW)
  Maintenance
  * Sevoflurane
  * Dexmedetomidine 0.4 mcg/kg/hr IV infusion using IBW (may titrate based on patient response between 0.3-0.5mcg/kg/hr)
  * Lidocaine 2mg/kg/hr IV infusion using IBW
  * May use esmolol as needed to treat SBP or HR > 20% of baseline
  * Neuromuscular blockade at the discretion of anesthesiology team
  Emergence
  * Dexmedetomidine infusion turned off during laparoscopic desufflation
  * Lidocaine infusion turned off at skin closure
  * Neuromuscular reversal, dosed according to VM protocol
  * Pt extubated and brought to PACU
  * PACU opioid orders per anesthesiology team
  Post-operative Nausea/Vomiting Prophylaxis
  -4mg dexamethasone, 1mg haloperidol, scopolamine patch
  Non Opioid Analgesics: see arm/group description
Period: Overall Study
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Started | 86 | 95
Completed | 86 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen | Total
Number analyzed (Participants) | 86 | 95 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.6) | 46.3 (13.1) | 46.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 74 | 144
  Male | 16 | 21 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Median (Inter-Quartile Range); unit: kilograms] | 124 [109 to 139] | 122 [106 to 138] | 123 [108 to 138]
Ideal Body Weight (IBW) [Median (Inter-Quartile Range); unit: kilograms] | 59 [53.5 to 64.5] | 60 [53.5 to 66.5] | 60 [54.5 to 65.5]
Body Mass Index [Median (Inter-Quartile Range); unit: kilograms/meter^2] | 44 [39 to 49] | 43 [38 to 48] | 43 [38 to 48]
American Society of Anesthesiologists (ASA) class [Count of Participants; unit: Participants] — ASA classification ranges from 1 - 6 based on a patient's preoperative comorbid conditions. ASA classification is a grading system used by anesthesiologists to assess a patient's health before surgery. The system assigns a patient a score from ASA 1 to ASA 6, with higher numbers indicating a higher risk of complications. The ASA classification system is used in conjunction with other factors, such as the type of surgery, to help predict the risk of surgery.
  Participants
    2 | 30 | 16 | 46
    3 | 56 | 79 | 135

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Opioid Consumption
Description: Total amount of opioid use within the first 24 hours after surgery in mg of oral morphine equivalent doses
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg oral morphine equivalents (OMEs)
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 86 | 95
mg oral morphine equivalents (OMEs)
  Including PACU | 51 (34) | 55 (31)
  Excluding PACU | 27 (24) | 32 (23)

2. Secondary Outcome: Length of Time Under General Anesthesia
Description: Time from induction to emergence of anesthesia
Time Frame: 1-5 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 86 | 95
hours | 3.47 (1.02) | 3.32 (1.04)

3. Secondary Outcome: Percentage of Patients With Opioid-related Adverse Effects
Description: Adverse effects include postoperative nausea, vomiting, pruritis, and respiratory depression. Some subjective, patient-reported data collection failed; these participants were excluded from this outcome.
Time Frame: 24 hours
Population: Some subjective, patient-reported data collection failed; these participants were excluded from this outcome
Measure: Count of Participants; unit: Participants
Groups:
- Control Group A- Opioid-based Regimen: Preop - Multimodals unless contraindicated
  Induction
  Fentanyl (50mcg IV) Lidocaine 1.5mg/kg IV bolus using IBW (Ideal body weight) Propofol 2-3mg/kg IV bolus Neuromuscular blockade per Anesthesiology team discretion Maintenance
  Sevoflurane Neuromuscular blockade at discretion of anesthesiology team May use fentanyl to treat SBP or HR > 20% of baseline Emergence
  Neuromuscular reversal, dosed according to Virginia Mason protocol May titrate fentanyl per anesthesiology team throughout the case. Patient extubated and brought to PACU PACU opioid orders per anesthesiology team
  Post-operative Nausea/Vomiting Prophylaxis
  -4mg dexamethasone, 1mg haloperidol, scopolamine patch
  Opioid Anesthetics: see arm/group description
- Experimental Group B- Opioid-free Regimen: Preop - Multimodals unless contraindicated
  Induction
  Dexmedetomidine 1mcg/kg IV bolus over 10 minutes using IBW Lidocaine 1.5mg/kg IV bolus using IBW Propofol 2-3mg/kg IV bolus Neuromuscular blockade per Anesthesiology team discretion Ketamine 0.5mg/kg IV bolus (based on IBW) Maintenance
  Sevoflurane Dexmedetomidine 0.4 mcg/kg/hr IV infusion using IBW (may titrate based on patient response between 0.3-0.5mcg/kg/hr) Lidocaine 2mg/kg/hr IV infusion using IBW May use esmolol as needed to treat SBP or HR > 20% of baseline Neuromuscular blockade at the discretion of anesthesiology team Emergence
  Dexmedetomidine infusion turned off during laparoscopic desufflation Lidocaine infusion turned off at skin closure Neuromuscular reversal, dosed according to VM protocol Pt extubated and brought to PACU PACU opioid orders per anesthesiology team Post-operative Nausea/Vomiting Prophylaxis
  -4mg dexamethasone, 1mg haloperidol, scopolamine patch
  Non Opioid Analgesics: see arm/group description
Arm/Group | Control Group A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 86 | 95
Participants
  Experienced vomiting: number analyzed (Participants) | 80 | 86
  Experienced vomiting | 19 | 16
  Experienced pruritis: number analyzed (Participants) | 80 | 86
  Experienced pruritis | 2 | 4
  Oxygen requirement beyond postanesthesia care unit: number analyzed (Participants) | 80 | 87
  Oxygen requirement beyond postanesthesia care unit | 21 | 29

4. Secondary Outcome: Length of Time to Recover From General Anesthesia
Description: Time from arrival to PACU to "ready for PACU discharge"
Time Frame: 1-3 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 86 | 95
hours | 1.33 (0.62) | 1.41 (0.75)

5. Secondary Outcome: Length of Hospital Stay
Description: Time from PACU arrival to discharge date and time in days
Time Frame: 1-5 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 86 | 95
days | 1.45 (0.6) | 1.58 (0.76)

6. Secondary Outcome: Overall Patient Satisfaction With Analgesia: Yes or no
Description: Number of Participants With Overall Patient Satisfaction With Analgesia
Time Frame: 24 hours
Population: Some subjective, patient-reported data collection failed; these participants were excluded from this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 80 | 87
Participants | 73 | 72

7. Secondary Outcome: Number of Participants With Post-surgical Opioid Prescription Refills up to 30 Days
Description: Number of participates with opioid prescription refills since surgery within 30 day after surgery
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 86 | 95
Participants | 9 | 10

8. Secondary Outcome: Percentage of Patients Treated for General Anesthetic Adverse Effects
Description: Episodes of severe bradycardia or treated hypotension intraoperatively
Time Frame: Intraoperative, between time entering OR and PACU arrival time
Population: Lowest intra-op heart rate less than 50 beats per minute
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 86 | 95
Participants
  Severe bradycardia intraoperatively (lowest HR <50 bpm) | 10 | 17
  Received phenylephrine intraoperatively | 41 | 67
  Received ephedrine intraoperatively | 28 | 54

9. Secondary Outcome: Number of Participants With Post-surgical Opioid Prescription Refills Between 30 Days to 3 Months After Surgery
Description: Number of participates with opioid prescription refills since surgery between 30 day and 3 months after surgery
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
Number analyzed (Participants) | 86 | 95
Participants | 8 | 4

ADVERSE EVENTS:
Time Frame: 3 months
Description: Some subjective, patient-reported data collection failed; these participants were excluded from these outcome.
Arm/Group | Control Goup A- Opioid-based Regimen | Experimental Group B- Opioid-free Regimen
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/95
Other Adverse Events (participants affected / at risk) | 51/86 | 62/95
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Control Goup A- Opioid-based Regimen (N=86) | Experimental Group B- Opioid-free Regimen (N=95)
Oxygen requirement beyond postanesthesia care unit (Respiratory, thoracic and mediastinal disorders) | 21/80 (21) | 29/87 (29)
Experienced vomiting (Gastrointestinal disorders) | 19/80 (19) | 16/86 (16)
Experienced pruritis (Skin and subcutaneous tissue disorders) | 2/80 (2) | 4/86 (4)
Severe bradycardia (Cardiac disorders) | 10 (10) | 17 (17) — Intraoperative heart rate less than 50 beats per minute
Experienced sedation beyond postanesthesia care unit (Nervous system disorders) | 25/80 (25) | 21/87 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04081545/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04081545/ICF_001.pdf